CLINICAL TRIAL: NCT02656771
Title: Evaluation of Uncemented Echo Bi-Metric Full Proximal Profile THA Stem Versus Uncemented Bi-Metric Porous Primary THA Stem in a Randomized Controlled Trial Using RSA and DXA
Brief Title: Evaluation of Stability of Two Uncemented Hip Implants Used for Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other); Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Karen Dyreborg, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THA1-KD-14
Record Dates: First submitted 2016-01-13; First posted 2016-01-15 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Osteoarthritis, Hip
Keywords: THA; Hip; arthroplasties
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Echo Bi-Metric THA stem (Active Comparator): Uncemented titanium alloy press-fit stem with a proximal plasma spray porous titanium coating designed for bone ingrowth and the distal part of the stem has a roughened titanium surface for bone on-growth.
  It is a relatively new implant that is now in routine clinical use. The stem uses many of the features of the known and used Integral® and Bi-Metric® hip stems while integrating new design features to further enhance clinical performance such as a reduced neck geometry to allow for increased ROM and decreased risk of neck impingement, a polished neck designed to reduce debris should impingement occur and a polished bullet-shape distal tip to reduce distal stresses.
  Interventions: Device: Echo Bi-Metric
- Bi-Metric Porous Primary THA stem (No Intervention): Uncemented titanium alloy press-fit stem with a proximal plasma spray porous titanium coating designed for bone ingrowth and the distal part of the stem has a roughened titanium surface for bone on-growth.
  It was introduced in 1984 and have shown good clinical results and excellent stem survival in register studies

INTERVENTIONS:
Device: Echo Bi-Metric — The insertion of the Echo® Bi-Metric® THA stem
  Arms: Echo Bi-Metric THA stem

SUMMARY:
The purpose of this study is to measure quantitatively the implant stability and implant related remodeling of the periprosthetic femoral bone of the new uncemented Echo® Bi-Metric® Full proximal Profile total hip arthroplasty (THA) stem, and compare it to the classical uncemented Bi-Metric® Porous Primary THA stem by measuring migration of the stem assessed by model-based radiosteriometric analysis (MB-RSA) and measuring the periprosthetic adaptive bone remodeling assessed by dual-energy x-ray absorptiometry (DXA).

DETAILED DESCRIPTION:
Material and Methods Hypothesis The uncemented Echo® Bi-Metric® Full proximal Profile THA stem shows less migration and less bone loss of the periprosthetic bone compared to the uncemented Bi-Metric® Porous Primary THA stem.

Operation All operations will be performed by 4 experienced hip surgeons from the Hip unit at the Department of Orthopedic Surgery, Gentofte Hospital, Gentofte, Denmark. Each of the surgeons performs approximately 120 THA-operations a year.

Surgery is performed according to a standard procedure with a postero-lateral approach and following the manufacturers' recommendations. During surgery a minimum of 4 Tantalum markers (0.8mm) are inserted in the bone of the proximal femur for defining the bone segment in the RSA analysis. All patients receive the same uncemented hemispheric acetabular cup (Exceed) with a highly cross-linked polyethylene liner. No local analgesic is injected. Physiotherapy begins on the day of surgery and the patients will be mobilized with full weight-bearing using crutches. All patients will get oral anticoagulants according to praxis of the department (Xarelto until discharge), and prophylactic antibiotics (Dicloxacillin, 2 g preoperatively and 1g x 2 postoperatively) during the first 24 hours.

Research plan

1. Clinical examination performed preoperatively and with follow-up after 1 and 2 years with evaluation of the hip function using the Harris Hip Score (HHS); HHS is a questionnaire in which the patients reveal their level of pain, function, mobility and range of motion.
2. Conventional X-rays: To evaluate possible aseptic loosening, all patients will have a standardized full pelvic antero-posterior X-ray and a lateral X-ray with fixed magnification both preoperatively, postoperatively, at the 2 years follow-up visit and at the 5 years follow-up visit. Radiolucent lines at the bone-implant interface and evidence of osteolysis will be measured on both recordings. The standard Gruen zones will be used to record radiolucency surrounding the femoral component and the acetabular zones described by DeLee and Charnley will be used to record radiolucency surrounding the acetabular component. The apparent thickness of the radiolucency within these zones will be recorded. Evidence of osteolysis (radiolucency >2mm thickness) in the periprosthetic tissue of the acetabular or femoral component will be considered a failure.
3. DXA analysis of the changes in BMD of the periprosthetic Gruen zones will be used to evaluate the adaptive bone remodeling after the implantation of the two different stems. DXA analysis will be performed preoperatively of the hip and proximal tibia as baseline, then again within the first postoperative week and subsequently at 3 months, 6 months, 1 year, 2 years and 5 years. The precision of the BMD measurements of the proximal femur will be estimated from double measurements of patients (n=12) included in the study.
4. MB-RSA measurements of migration of the femoral component. A MB-RSA system will be used; a technique in which the position of the prosthesis is assessed by matching a virtual projection of a 3D-model of the prosthesis to the actual radiographic projection. It does not require former times' special implants with attached markers. The patients will be x-rayed within the first postoperative week and subsequently at 3 months, 6 months, 1 year, 2 years and 5 years using 2 fixed X-ray tubes with the patient in supine position and a uniplanar calibration cage will be used. The precision of the measurements of migration will be estimated from sets of double X-rays of patients (n=12) included in the study.
5. Patient reported outcome measurements. It is planned also to ask the patients preoperatively and after 6, 12 and 24 months to do a patient-reported outcome measurement using the Oxford Hip Score (OHS).
6. Long term follow-up. 5-year follow-up including all above mentioned parameters will be performed.

Calculations of sample size Migration (RSA). Several published RSA studies are available but none evaluating an uncemented Bi-Metric stem including data for the most clinically relevant migration between 1 and 2 years. Quite a lot of RSA studies evaluating migration of both cemented and uncemented femoral stems have been published, but most investigators give the variability of their RSA results as total range or standard error of mean. We have decided for our sample size calculation to use the average standard deviation (SD) -for the migration after 2 years of follow-up from two previously published studies (including data from one uncemented (n=22) and two cemented stems (n=82), where clear information regarding SD was available in the publication.

Investigators performed the calculation using the parameter MTPM two years postoperatively using:

Type I error = 5% Type II error = 15 % MIREDIF = 0.6 mm SD = 0.69 mm Calculation resulted in a sample size of n = 23 in each group.

Bone remodeling (DXA). The expected prospective decrease in BMD of the proximal femur after insertion of an uncemented THA is most pronounced in Gruen zones 1 and 7 with decreases of respectively 13-21% and 10-31%. In this study investigator intend to measure a significant difference (MIREDIF) in percentage changes in BMD between the two groups of 7.5%. Even though several studies evaluating prospective changes in BMD around a femoral stem have been published, investigator did not find a study with precise information of the SD of the percentages in BMD. Thus, investigator estimated a SD of the changes in BMD of 8% that could be used for calculating sample size in our study.

Using:

Type I error = 5% Type II error = 15% and MIREDIF = 7.5% SD = 8% Calculation resulted in a sample size of n = 20 in each group. Based upon the above sample size calculations for both RSA and DXA investigator have planned to include and randomize a total of: 60 patients.

This will secure a high statistical power of the study (even if some of the participants should drop out during the study) that can be kept even if the study is continued beyond 2 years of follow-up.

Randomization Allocation to the Echo® Bi-Metric® group or control group (Bi-Metric® group) is performed on a random basis (block randomization with 10 in each block). Randomization is done on the day of surgery with a closed non-transparent envelope opened in the operation theatre when the patient is ready for surgery.

Due to visual difference of the two prostheses, the surgeon and personnel present will know which of the prostheses the patient shall receive.

Ethical considerations This investigation will be performed in accordance with the principles of the Helsinki Declaration, and all patients will receive both oral and written information before informed consent to participate is obtained. It will be the investigators job to inform all patients until they completely understand all aspects of participation. At any time being the patient will be able to cancel participation (also without any explanation) in this investigation. The patient will receive the best possible treatment in any circumstance.

The study will not be started until approval from the Scientific Ethical Committee of the Capital Region of Denmark and the Danish Data Protection Agency has been obtained, and it will be registered at clinicaltrials.gov.

We do not expect the patients participating in the study to experience any specific side effects or complications related directly to the use of the two orthopedic implants. A potential difference between the two prostheses is expected only to be measurable using very precise techniques such as DXA and RSA.

Radiation dose to the patients from both RSA and DXA is low compared with conventional x-ray examinations. The total accumulated radiation dose to a patient participating in all examinations during the study is estimated to be approximately 0.1 mSv.

Tantalum has been used for more than 50 years and is a very biocompatible material. Tantalum beads for RSA have been used especially in Sweden in several clinical studies for more than 20 years. More than 20.000 beads have been implanted in more than 2.000 patients and no side effects from Tantalum beads have been observed.

Risks and inconveniences There will always be risks associated with operation. This investigation will not add to the general risks of getting THA. Patients participating must accept some inconvenience in terms of additional examinations and hence transportation to and from the hospitals.

Adverse events Adverse events are defined as any harmful and unwanted event, sign or symptom to occur in relation to this trial. All adverse events will be recorded in the CRF and will include details concerning the nature, onset, duration, severity, relationship to the device and relationship to the operative procedure and outcome. The affected patient(s) will be questioned about any adverse event(s) at each subsequent follow-up visit.

Patients experiencing adverse events will be relevantly monitored by clinical assessment and lab examinations decided by the treating physician. All adverse events will be monitored until recovery or stabilization.

Information and consent Patients who are planned to receive a THA (and fits within the inclusion and exclusion criteria of the study) at Gentofte Hospital will be informed about the trial in the preoperative interview. In addition to the oral information provided, the patients will be given written information. This conversation will take place in an enclosed space without distractions or interruptions. The patient will receive adequate verbal and written information about the purposes, processes, potential benefits and risks including possible side effects. Investigator will ensure all patients have read and understood the information and consent form. Patients will be informed that they are entitled to consideration before consent is given. The subjects will also be informed that it is voluntary and that they at any time may withdraw from the trial. It is the investigator's responsibility to ensure the above.

There will be obtained written informed consent from all subjects before enrollment, and a copy of the information and consent form will be given to the subjects.

Existing legislations made by the Scientific Ethical Committee regarding informed consent will be followed.

Data protection All information will be kept confidential, and all data handled according the guidelines of the Danish Data Protection agency. The persons involved in this trial are obliged to professional secrecy. The investigator will maintain a list of identification of all enrolled patients. This list will contain the patients' full names and dates of birth (including social security numbers (CPR-numbers)).

Collected data will be recorded in a case report form (CRF). CRFs and the medical records will be made available to third parties according to Danish law. Patients will be informed in writing that the results will be stored and analyzed in a computer which preserve patients' anonymity and that the local laws regarding personal data will be complied.

Patients will also receive written information concerning the possibility of audit from the public authorities, and patients will be informed that the GCP unit of Copenhagen University Hospital likewise is granted access.

Investigator ensures that the project will follow the rules of Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients bound to undergo total hip arthroplasty at the Department of Orthopedic - Surgery, Gentofte Hospital, Denmark.
* Patients who have consented in writing to participate after having understood what it entails.
* Patients diagnosed with primary osteoarthritis of one or both hips.

Exclusion Criteria:

* Infection including osteomyelitis and sepsis.
* Exclusion as a result of technical shortcomings such as poor image quality, estimated by the investigator.
* Diseases affecting the bone metabolism (osteoporosis, Pagets disease, hyperparathyreoidism etc.).
* Uncooperative patient or patients with neurological disorders who are considered incapable of following directions.
* Patients with alcohol or drug abuse, estimated by the investigators.
* Patients considered unable to understand the information in patients-papers, or who do not want to participate in the study.
* Patients who do not speak nor understand Danish.
* Pregnancy

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-01; Primary Completion 2019-07 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Migration of the stem | 2 years
  The differences between the two stem designs are evaluated by measurements of migration of the stem assesed by Radiosteriometric analysis (RSA)

SECONDARY OUTCOMES:
Adaptive bone remodeling | 2 years
  The differences of the two stems are evaluated by measurements of the adaptive bone remodeling of the periprostetic area (femur) assesed by dual energy X-ray absorptiometry (DXA)
Hip function | 2 years
  Hip function postoperatively assesed by Harris Hip Score and Oxford Hip Score

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Petersen, Professor, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Gentofte Hospital, Hellerup, Denmark

REFERENCES:
- [Background] Haugan K, Husby OS, Klaksvik J, Foss OA. The migration pattern of the Charnley femoral stem: a five-year follow-up RSA study in a well-functioning patient group. J Orthop Traumatol. 2012 Sep;13(3):137-43. doi: 10.1007/s10195-012-0187-x. Epub 2012 May 11. PMID 22576838
- [Background] Nieuwenhuijse MJ, Valstar ER, Kaptein BL, Nelissen RG. Good diagnostic performance of early migration as a predictor of late aseptic loosening of acetabular cups: results from ten years of follow-up with Roentgen stereophotogrammetric analysis (RSA). J Bone Joint Surg Am. 2012 May 16;94(10):874-80. doi: 10.2106/JBJS.K.00305. PMID 22617914
- [Background] O'Neill SC, Queally JM, Devitt BM, Doran PP, O'Byrne JM. The role of osteoblasts in peri-prosthetic osteolysis. Bone Joint J. 2013 Aug;95-B(8):1022-6. doi: 10.1302/0301-620X.95B8.31229. PMID 23908414
- [Background] Jiang Y, Jia T, Wooley PH, Yang SY. Current research in the pathogenesis of aseptic implant loosening associated with particulate wear debris. Acta Orthop Belg. 2013 Feb;79(1):1-9. PMID 23547507
- [Background] Nelissen RG, Pijls BG, Karrholm J, Malchau H, Nieuwenhuijse MJ, Valstar ER. RSA and registries: the quest for phased introduction of new implants. J Bone Joint Surg Am. 2011 Dec 21;93 Suppl 3:62-5. doi: 10.2106/JBJS.K.00907. PMID 22262426
- [Background] Selvik G. Roentgen stereophotogrammetry. A method for the study of the kinematics of the skeletal system. Acta Orthop Scand Suppl. 1989;232:1-51. PMID 2686344
- [Background] Ryd L. Micromotion in knee arthroplasty. A roentgen stereophotogrammetric analysis of tibial component fixation. Acta Orthop Scand Suppl. 1986;220:1-80. PMID 3461667
- [Background] Snorrason F, Karrholm J. Primary migration of fully-threaded acetabular prostheses. A roentgen stereophotogrammetric analysis. J Bone Joint Surg Br. 1990 Jul;72(4):647-52. doi: 10.1302/0301-620X.72B4.2199453.
- [Background] Stiehl JB. Early cup instability with RSA predicts long-term aseptic loosening: commentary on an article by Marc J. Nieuwenhuijse, BSc, MD, et al.: "Good diagnostic performance of early migration as a predictor of late aseptic loosening of acetabular cups. Results from ten years of follow-up with Roentgen stereophotogrammetric analysis (RSA)". J Bone Joint Surg Am. 2012 May 16;94(10):e70. doi: 10.2106/JBJS.L.00080. No abstract available. PMID 22617936
- See also: Danish Hip Arthroplasty Registry, annual report 2012 — http://www.dhr.dk/Ny%20mappe/rapporter/DHR%20årsrapport%202012%20final-29.8.2012.pdf